CLINICAL TRIAL: NCT04486586
Title: Effects of Transcranial Direct Current Stimulation in Primary Progressive Aphasia (PPA)
Brief Title: Effects of tDCS on Apraxia of Speech in Non-Fluent Primary Progressive Aphasia
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: The study was withdrawn due to a shift in research priorities, with the decision made to focus resources on other studies that align more closely with the current strategic goals.
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: NA_00071337-2
Record Dates: First submitted 2020-07-20; First posted 2020-07-24 (Actual); Last update posted 2025-04-24 (Actual); Status verified 2025-04

CONDITIONS: Primary Progressive Aphasia
Keywords: transcranial direct current stimulation (tDCS); neurodegeneration; language therapy; primary progressive aphasia (PPA); apraxia of speech (AOS)
MeSH Terms: conditions — Aphasia, Primary Progressive; Nerve Degeneration; Apraxias | interventions — Speech Therapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Active tDCS plus Speech-Language Therapy first (Experimental): Active tDCS will be applied at the beginning of 45 minutes speech-language therapy session and then participant will be switched to sham tDCS after a washout period.
  Interventions: Device: Active tDCS plus Speech-Language Therapy; Device: Sham plus Speech-Language Therapy
- Sham plus Speech-Language Therapy first (Sham Comparator): Sham will be applied at the beginning of 45 minutes speech-language therapy session and then participant will be switched to an active tDCS after a washout period.
  Interventions: Device: Active tDCS plus Speech-Language Therapy; Device: Sham plus Speech-Language Therapy

INTERVENTIONS:
Device: Active tDCS plus Speech-Language Therapy — Stimulation will be delivered by a battery-driven constant current stimulator. The electrical current will be administered to a pre-specified region of the brain (inferior frontal gyrus). The stimulation will be delivered at an intensity of 2 mA (estimated current density 0.04 mA/cm^2; estimated total charge 0.048 C/cm^2) in a ramp-like fashion for a maximum of 20 minutes. Speech-language therapy will target apraxia of speech (AOS).
Device: Sham plus Speech-Language Therapy — Speech-language therapy will be administered during sham stimulation. Current will be administered in a ramp-line fashion but after the ramping the intensity will drop to 0 mA. Speech-language therapy will target apraxia of speech (AOS).

SUMMARY:
Primary progressive aphasia (PPA) is a neurodegenerative disease that affects first and foremost language abilities. There are three different variants of PPA, each a relatively distinct speech and language profile. For individuals with non-fluent variant PPA (nfvPPA), a core symptom is apraxia of speech (AOS), which is defined as an oral motor speech disorder. Such a disorder inhibits one's ability to translate speech plans into motor plans and results in longer segmental durations and reduced rate of syllabic production.

This research project investigates the behavioral and neuromodulatory effects of transcranial direct current stimulation (tDCS) during language therapy in participants with nfvPPA over time. Anodal tDCS targeting the left inferior frontal gyrus (IFG) administered in combination with language therapy is expected to be more beneficial when compared to language therapy alone (sham). The investigators believe tDCS during language therapy will 1) improve language performance or decrease rate of decline, 2) promote better-sustained effects at 2 weeks and 2 months post-treatment, and 3) produce generalization to untrained language items and some other cognitive functions. Resting-state fMRI, diffusion tensor imaging (DTI), and volumetric data are also collected to investigate changes in functional brain connectivity associated with tDCS in individuals with PPA.

A better understanding of the therapeutic and neuromodulatory mechanisms of tDCS as an adjunct to language therapy in nfvPPA may have a significant impact on the development of effective therapies for PPA, and may offer insight into ways of impeding neurodegeneration that may improve patients' quality of life, as well as extend patients' ability to work and manage patients' affairs.

DETAILED DESCRIPTION:
A. Evaluation Tasks

Language Tasks:

Participants will be administered baseline language and cognitive tasks, including 1 or more of the following, depending on participants' residual language and cognitive skills:

a) writing to dictation b) oral spelling c) oral and written naming of pictures d) word-picture matching f) written and oral picture description g) digit span h) spatial span i) verbal learning j) grammatical sentence production k) oral word repetition l) sentence comprehension

Quality of Life questionnaires:

Participants will be administered standardized and non-standardized quality-of-life questionnaires before, after, and at follow-up intervals of each experimental period. The purpose of these questionnaires is to assess whether the proposed interventions have affected participants' well-being and the general quality of participants' life.

B. AOS Intervention

Intervention involves oral word repetition of increasingly complex words. The goal is to improve volitional control of participants' articulators in order to produce co-articulated, intelligible speech, as well as improve prosody, voice quality, and speech fluency.

C. Assessment of Language Therapy Tasks:

Follow-up assessments will probe all sets of increasingly complex words targeted in intervention and as well as word sets not targeted in intervention to assess near-transfer generalization. Other language and cognitive tasks will be assessed for far-transfer generalization. Differences in baseline measures in pre- and post-intervention accuracy for word production for each patient will be evaluated using the following: percentages of total number of words correct, arithmetic differences between percentage scores, and permutation tests (Pearson's chi-square test; Fisher's exact test).

C. tDCS Methods:

Participants will take part in 10-15 consecutive training sessions (3-5 per week), separated by 2 months. Anodal tDCS has typically been shown to up-regulate neuronal excitability and produce enhancement of behavioral performance. A Soterix-CT device will be delivering current at an intensity of 1-2 mA (estimated current density 0.04 mA/cm^2; estimated total charge 0.048 C/cm^2) for a maximum of 20 minutes in the tDCS groups and for a maximum of 30 seconds in the Sham group. For both interventions (tDCS and Sham) the electrical current will be increased in a ramp-like fashion at the onset of the stimulation eliciting a transient tingling sensation on the scalp that usually disappears over seconds.

D. Imaging Methods:

Imaging will be performed at the beginning of enrollment, before and after each 12-to-15-day tDCS treatment, and at follow-up intervals for up to 8 time points per individual on a 3T Philips system, and will consist of resting-state fMRI (rsfMRI), MPRAGE, and diffusion tensor imaging (DTI). Each scanning session will last approximately 1 hour.

E. Statistical Analyses:

In the within-subject crossover protocol, each participant will be administered two experimental conditions: IFG tDCS+language (tDCS intervention) and IFG sham+language (sham treatment). All analyses, behavioral and imaging, will be under the oversight of the study statisticians.

F. Study duration and number of study visits required of research participants.

Before any intervention, participants will be randomly assigned to either sham or tDCS experimental conditions. After 1-3 weeks of tDCS application (3-5 sessions in a week, 10-15 sessions per stimulation site) there will be an interval of approximately 2 months and then the investigators will implement the other two tDCS conditions in a within-subject cross-over design. Participants will be followed-up at 2-week and 2-month follow-up intervals.

G. Blinding, including justification for blinding or not blinding the trial, if applicable.

Participants will be blinded to the application of anodal or sham tDCS. To achieve blinding, all participants will be fitted with the tDCS electrodes placed over the left inferior frontal gyrus (IFG). The Soterix-CT device will be used for double-blinding purposes.

H. Justification of why participants will not receive routine care or will have current therapy stopped

Participation in this study will not disrupt any current care or therapy.

I. Justification for inclusion of a placebo or non-treatment group

All participants will undergo active and sham conditions, thus serving as participants' own control.

J. Definition of treatment failure or participant removal criteria

Participants will be removed from the study if participants are unable to comply with task instructions or tolerate the tDCS procedure.

K. Description of what happens to participants receiving therapy when study ends or if a participant's participation in the study ends prematurely

When the study ends participants will continue to receive management with participants' neurologist as usual. If a patient's participation in the study ends prematurely s/he will still receive care as before. In sum, termination of the study or termination of participation in it will not affect regular therapy he or she may be receiving.

L. Qualification of investigators:

The principal investigator (PI) and co-investigators have extensive research and clinical experience with all study tasks: behavioral language therapy (including AOS intervention). The investigators have already published tDCS studies showing positive results in spelling.

ELIGIBILITY:
Inclusion Criteria:

* Must be clinically diagnosed with nfvPPA or unclassifiable PPA. Diagnosis will be based on neuropsychological testing, language testing (most commonly the Western Aphasia Battery), MRI and clinical assessment.
* Must be right-handed.
* Must be speaker of English.
* Must have at least 9th grade education.

Exclusion Criteria:

* Uncorrected visual or hearing impairment by self report.
* Stroke/other premorbid neurological disorder affecting the brain.
* Any other language-based learning disorder other than PPA.
* Inability to follow directions for baseline tasks.
* Western Aphasia Battery Aphasia Quotient (AQ) <30 (indicating severe language impairment).

Exclusion Criteria for MRI Participation:

* Severe claustrophobia.
* Cardiac pacemakers or ferromagnetic implants.
* Pregnant women.

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2013-04 (Actual); Primary Completion 2025-04 (Estimated); Study Completion 2025-04 (Estimated)

PRIMARY OUTCOMES:
Change in segmental duration of vowels of trained words | Before intervention, immediately after intervention, 2 weeks post intervention and 2 months post intervention
  Duration of vowels for trained words (practiced in therapy) will be measured in milliseconds (ms) via acoustic analyses. Investigators will compute the change in outcome over time: before intervention versus each time point after. Decrease in duration is considered a benefit.
Change in segmental duration of vowels of untrained words | Before intervention, immediately after intervention, 2 weeks post intervention and 2 months post intervention
  Duration of vowels for untrained words (not practiced in therapy) will be measured in milliseconds (ms) via acoustic analyses. Investigators will compute the change in outcome over time: before intervention versus each time point after. Decrease in duration is considered a benefit.
Change in segmental duration of consonants of trained words | Before intervention, immediately after intervention, 2 weeks post intervention and 2 months post intervention
  Duration of consonants for trained words (practiced in therapy) will be measured in milliseconds (ms) via acoustic analyses. Investigators will compute the change in outcome over time: before intervention versus each time point after. Decrease in duration is considered a benefit.
Change in segmental duration of consonants of untrained words | Before intervention, immediately after intervention, 2 weeks post intervention and 2 months post intervention
  Duration of consonants for untrained words (not practiced in therapy) will be measured in milliseconds (ms) via acoustic analyses. Investigators will compute the change in outcome over time: before intervention versus each time point after. Decrease in duration is considered a benefit.
Change in speech fluency on trained words | Before intervention, immediately after intervention, 2 weeks post intervention and 2 months post intervention
  Speech fluency will be measured on trained words (practiced in therapy) using the mean log of sound duration collected via acoustic analyses. Investigators will compute the change in outcome over time: before intervention versus each time point after. Lower log duration indicates faster speech production. A decrease in sound duration is considered a benefit.
Change in speech fluency on untrained words | Before intervention, immediately after intervention, 2 weeks post intervention and 2 months post intervention
  Speech fluency will be measured on untrained words (not practiced in therapy) using the mean log of sound duration collected via acoustic analyses. Investigators will compute the change in outcome over time: before intervention versus each time point after. Lower log duration indicates faster speech production. A decrease in sound duration is considered a benefit.

SECONDARY OUTCOMES:
Change in prosody/intonation of trained words | Before intervention, immediately after intervention, 2 weeks post intervention and 2 months post intervention
  Prosody/intonation for trained words (practiced in therapy) will be measured using mean fundamental frequency (F0), which is frequency at which vocal folds vibrate in voiced sounds. Such measurements will come from acoustic analyses. Investigators will compute the change in outcome over time: before intervention versus each time point after. Consistency over time is considered a benefit.
Change in prosody/intonation of untrained words | Before intervention, immediately after intervention, 2 weeks post intervention and 2 months post intervention
  Prosody/intonation for untrained words (not practiced in therapy) will be measured using mean fundamental frequency (f0), which is frequency at which vocal folds vibrate in voiced sounds. Such measurements will come from acoustic analyses. Investigators will compute the change in outcome over time: before intervention versus each time point after. Consistency over time is considered a benefit.
Change in syntactic comprehension as assessed by Subject-relative, Object-relative, Active, Passive (S.O.A.P.) Syntactic Battery | Before intervention, immediately after intervention, 2 weeks post intervention and 2 months post intervention
  The 40-item Subject-relative, Object-relative, Active, Passive (S.O.A.P.) Syntactic Battery of various sub-tests will be used to assess argument structure comprehension and production. The investigators will compute the raw score of items correct and transform to percent correct (range: 0-100). Subsequently, the investigators will compute change in outcome in percent difference between before intervention and each time point after. Increase in score is considered a benefit.
Change in verbal fluency task score | Before intervention, immediately after intervention, 2 weeks post intervention and 2 months post intervention
  Verbal fluency tasks (semantic and letter fluency) involve generating as many words as possible in one minute. Scoring will be based on number of words generated per minute. The investigators will compute the raw score of items correct and subsequently the percent difference between before intervention and each time point after. Increase in score is considered a benefit.
Change in semantic content of connected speech | Before intervention, immediately after intervention, 2 weeks post intervention and 2 months post intervention
  Using the Cookie Theft image from the Boston Diagnostic Aphasia Examination (BDAE) and the Circus image from the Apraxia Battery for Adults (ABA) investigators will obtain representative language samples as participants describe the images. The investigators will compute the raw score of items (semantics) correct and transform to percent correct (range: 0-100%), computing change in outcome in percent difference between before intervention and each time point after. Increase in score is considered a benefit.
Change in oral naming Boston Naming Test score | Before intervention, immediately after intervention, 2 weeks post intervention and 2 months post intervention
  The Boston Naming Test is a widely used picture naming test that detects lexical retrieval deficits in the oral modality. The investigators will compute the raw score of items correct and transform to percent correct (range: 0-100%), computing change in outcome in percent difference between before intervention and each time point after. Increase in score is considered a benefit.
Change in oral naming of action as assessed by Hopkins Assessment of Naming Actions (HANA) | Before intervention, immediately after intervention, 2 weeks post intervention and 2 months post intervention
  Accuracy in oral naming of actions will be assessed using HANA. The investigators will compute the raw score of items correct and transform to percent correct (range: 0-100%), computing change in outcome in percent difference between before intervention and each time point after. Increase in score is considered a benefit.
Change in digit span forward score | Before intervention, immediately after intervention, 2 weeks post intervention and 2 months post intervention
  Digit span forward involves the recall of a series of single digits (sets of 1-8 digits) in the same order the digits were presented. Scoring will be based on the number of consecutive digits correctly recalled. The investigators will compute the change in outcome between the time point before intervention and each time point after. Increase in score is considered a benefit.
Change in digit span backward score | Before intervention, immediately after intervention, 1 month post intervention and 3 months post intervention
  Digit span backward involves the recall of a series of single digits (sets of 1-8 digits) in the reverse order than the digits were presented. Scoring will be based on the number of consecutive digits correctly recalled. The investigators will compute the change in outcome between the time point before intervention and each time point after. Increase in score is considered a benefit.
Change in volumetric measurements of select brain regions | Before intervention, immediately after intervention and 3 months post intervention
  Using Magnetization-Prepared Rapid Gradient-Echo (MPRAGE) Magnetic Resonance Imaging (MRI) investigators will perform volumetric measurements of select brain regions. Measurements will be collected in millimeters cubed (mm^3).
Change in anisotropy of white matter tracts of select brain regions | Before intervention, immediately after intervention and 3 months post intervention
  Using Diffusion Weighted/Diffusion Tensor Imaging (DWI/DTI) investigators will estimate the anisotropy of the brain's white matter tracts on the brain regions of concern.
Change in location of white matter tracts of select brain regions | Before intervention, immediately after intervention and 3 months post intervention
  Using Diffusion Weighted/Diffusion Tensor Imaging (DWI/DTI) investigators will estimate the location of the brain's white matter tracts on the regions of concern.

CONTACTS AND LOCATIONS:
Overall Officials: Kyrana Tsapkini, PhD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Hospital, Baltimore, Maryland, United States